CLINICAL TRIAL: NCT02121249
Title: Randomized Comparative Trial of Minimally Invasive Robotic vs. Freehand in Short Adult Degenerative Spinal Fusion Surgeries
Brief Title: Clinical Trial of Minimally Invasive Robotic Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mazor_001
Record Dates: First submitted 2014-04-15; First posted 2014-04-23 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Degenerative Lumbar Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot assisted pedicle screw fixation (Experimental): posterior lumbar interbody fusion using Robot assisted pedicle screw fixation (Renaissance, Mazor Robotics Ltd, Caesare, Israel)
  Interventions: Device: Renaissance, Mazor Robotics Ltd, Caesare, Israel
- Free hand technique (Active Comparator): using Free hand technique, posterior lumbar interbody fusion (No specific device)
  Interventions: Procedure: free hand technique

INTERVENTIONS:
Device: Renaissance, Mazor Robotics Ltd, Caesare, Israel — Renaissance (Mazor Robotics Ltd, Caesare, Israel) is the name of the robot
  Other Names: (Renaissance, Mazor Robotics Ltd, Caesare, Israel)
  Arms: Robot assisted pedicle screw fixation
Procedure: free hand technique — No specific device is necessary in the "free hand technique"
  Arms: Free hand technique

SUMMARY:
The purpose of this study was to quantify potential short- and long-term benefits of robotically-guided minimally invasive spine surgery in instrumentation of degenerative lumbar or lumbosacral spine disease in adult patients, in comparison to instrumentation in a matching cohort of control patients performed using conventional freehand technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age from 40 years to 85 years), undergoing short (below 3 consecutive vertebrae) lumbar or lumbosacral fixation surgery.
* Primary surgery and revision surgery
* Patient capable of complying with study requirements
* Signed informed consent of patient or legal guardian

Exclusion Criteria:

* Infection or malignancy
* Primary abnormalities of bones (e.g. osteogenesis imperfecta)
* Primary muscle diseases, such as muscular dystrophy
* Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, neurofibroma)
* Spinal cord abnormalities with any neurologic symptoms or signs
* Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia
* Paraplegia
* Patients requiring anterior release or instrumentation
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
* Patient cannot follow study protocol, for any reason
* Patient (or legal guardian, when applicable) cannot or will not sign informed consent

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Pedicle screw instrumentation accuracy | within 7 days after operation
  The location of pedicle screw is evaluated by postoperative CTs in a subset of patients
Oswestry Disability Index | up to 5 year after operation, every year
  Health status

SECONDARY OUTCOMES:
Fusion rates | up to 5 year after operation
  This is assessed by postoperative computed tomography at 1 year after surgery
Operation duration | After operation
  Intraoperative time
intraoperative blood loss | after operation
  intraoperative blood loss
postoperative drainage | within 3 days after operation
  Total drainage after surgery
amount of transfusion | within 7 days after operation
  Total transfusion during and after surgery
time to ambulation | within 3 days after operation
  immediate postop to ambulation start
Change of Oswestry Disability Index | up to 5 year after surgery, every year
  Health status
Visual Analog Pain Scale | up to 5 year after operation, every year
  Pain status
SF-36 | up to 5 year after operation, every year
  Health status
Radiographic adjacent level degeneration | up to 5 year after operation, every year
  Radiographic changes according to UCLA, vertebral body translation, motion change, segmental kyphosis or lordosis, disc height changes

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Joong Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea